CLINICAL TRIAL: NCT03874052
Title: Phase I Study to Evaluate Safety of Ruxolitinib in Combination With Azacitidine + Venetoclax in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Ruxolitinib in Combination With Venetoclax With and Without Azacitidine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Saultz (Other)
Collaborators: AbbVie (Industry); Incyte Corporation (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Saultz, IND Holder, OHSU Knight Cancer Institute
Organization: OHSU Knight Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018238; NCI-2019-03272 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018238 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-01-10; First posted 2019-03-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Secondary Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Refractory Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Specimen Handling; Biopsy; ruxolitinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (ruxolitinib, venetoclax) (Experimental): Patients receive ruxolitinib PO BID and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive additional cycles of ruxolitinib and venetoclax at the discretion of the sponsor-investigator. Patients also undergo a skin punch biopsy and ECHO at screening and blood sample collection and bone marrow aspiration and biopsy throughout the study. (COMPLETE 04/04/2025)
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Procedure: Punch Biopsy; Other: Questionnaire Administration; Drug: Ruxolitinib; Drug: Venetoclax
- Arm 2 (ruxolitinib,venetoclax, azacitidine) (Experimental): Patients receive ruxolitinib PO BID, venetoclax PO QD, and azacitidine IV or SC on days 1-7 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO at screening and blood sample collection and bone marrow aspiration and biopsy throughout the study.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Procedure: Punch Biopsy; Other: Questionnaire Administration; Drug: Ruxolitinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm 2 (ruxolitinib,venetoclax, azacitidine)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Punch Biopsy — Undergo skin punch biopsy
  Other Names: BIOPSY, PUNCH; Punch Biopsy of Skin
Other: Questionnaire Administration — Ancillary studies
Drug: Ruxolitinib — Given PO
  Other Names: INCB 018424; INCB-018424; INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I trial studies the side effects and best dose of ruxolitinib when given together with venetoclax and compares the effect of ruxolitinib in combination with venetoclax to venetoclax and azacitidine in treating patients with acute myeloid leukemia (AML) that has come back (relapsed) or has not responded to treatment (refractory). Ruxolitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Azacitidine stops cells from making deoxyribonucleic acid and may kill cancer cells. It is a type of antimetabolite. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving ruxolitinib in combination with venetoclax and azacitidine may be safe, tolerable, and/or effective compare to ruxolitinib with venetoclax in treating patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate an maximum-tolerated dose (MTD) for ruxolitinib in combination with Ia. Venetoclax (Arm 1); Ib. Venetoclax and azacitidine (Arm 2).

SECONDARY OBJECTIVES:

I. To assess the efficacy of the study treatment. II. To assess the duration of clinical response. III. To assess the duration of clinical benefit. IV. To assess survival in the absence of treatment failure, hematologic relapse, or progressive disease.

V. To assess overall survival. VI. To assess overall acute toxicity and tolerability. VII. To assess the effect of ruxolitinib in combination with azacitidine + venetoclax on quality of life (QOL).

EXPLORATORY OBJECTIVES:

I. To assess in vitro kinase inhibitor sensitivity using participants' bone marrow (or peripheral blood).

II. To characterize changes in disease using molecular techniques (potentially including next-generation sequencing and/or BH3 profiling).

III. To assess the impact of changes in molecular disease features. IV. To determine the in vivo pharmacokinetics (PK)/pharmacodynamics (PD) parameters of the study drugs (Arm 1 only).

OUTLINE: This is a dose-escalation study of ruxolitinib in combination with fixed dose venetoclax with and without azacitdine. Patients are assigned to 1 of 2 arms.

ARM 1 (COMPLETE 04/04/2025): Patients receive ruxolitinib orally (PO) twice daily (BID) and venetoclax PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive additional cycles of ruxolitinib and venetoclax at the discretion of the sponsor-investigator. Patients also undergo a skin punch biopsy and echocardiography (ECHO) at screening and blood sample collection and bone marrow aspiration and biopsy throughout the study.

ARM 2: Patients receive ruxolitinib PO BID, venetoclax PO QD, and azacitidine intravenously (IV) or subcutaneously (SC) on days 1-7 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO at screening and blood sample collection and bone marrow aspiration and biopsy throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Age >= 18 years at time of informed consent. Persons of all genders and gender identities, and members of all races and ethnic groups will be included
* Morphologically documented relapsed/refractory (R/R) AML or R/R secondary AML (sAML) that has progressed after at least 1 prior therapy for AML

  * Prior treatment with venetoclax and azacitidine is allowed
  * Treatment with hydroxyurea will not be considered a line of therapy
  * Patients with morphologically documented myelodysplastic syndrome (MDS) that has progressed on hypomethylating agent (HMA) therapy also will be considered if the patient is ineligible for induction with intensive chemotherapy (IC), defined for this study as meeting one or more of the following criteria:

    * Severe cardiac disorder (e.g., congestive heart failure requiring treatment, left ventricular ejection fraction (LVEF) of ≤ 50%, or chronic stable angina)
    * Severe pulmonary disorder, certified by the managing physician
    * Creatinine clearance of < 45 ml/min or
    * Hepatic disorder with total bilirubin > 1.5 x upper limit of normal (ULN)
    * Eastern Cooperative Oncology Group (ECOG) equal to 2
    * Other comorbidity(ies) judged to be incompatible with high dose chemotherapy by the managing physician will be considered, at the discretion of the principal investigator (PI)
* ECOG performance status 0 to 2
* Persons of childbearing potential (PCBP) must have a negative serum or urine pregnancy test within 14 days prior to start of study drug administration
* Patients must agree to use an adequate method of contraception while on study treatment and for 120 days after the last dose of ruxolitinib for Arm 1 and 6 months after the last dose of azacitidine for Arm 2
* Must be able to take and absorb oral medications
* Creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hour urine collection
* Total serum bilirubin ≤ 1.5 x ULN unless thought to be due to leukemic involvement
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 3.0 x ULN unless thought to be due to leukemic involvement

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL or AML M3 subtype)
* Active central nervous system involvement with AML
* Currently receiving chemotherapy or investigational agents within or 5 half lives, or less of the planned start of treatment, with the exception of hydroxyurea for cytoreduction of proliferative disease
* Concurrent active malignancy with expected survival of less than 1 year, at the discretion of the investigator. For example, candidates with treated skin cancers, prostate cancer, breast cancer, etc. without metastatic disease are candidates for therapy since their expected survival exceeds that of relapsed or refractory AML
* Clinically significant graft versus host disease (GVHD) or active GVHD requiring initiation or escalation of treatment within 28-day screening period
* Participants with rapidly progressive disease (defined by blast count doubles within 48 hours) or organ dysfunction
* Documented cardiac insufficiency (e.g., symptomatic heart failure, left ventricular ejection fraction of ≤ 40%)
* Symptomatic shortness of breath or patient requires supplemental oxygen support
* Clinically significant coagulation abnormality, such as disseminated intravascular coagulation
* Known history of cerebrovascular accident, myocardial infarction, or intracranial hemorrhage within 2 months of enrollment
* Known clinically significant liver disease defined as ongoing drug-induced liver injury, chronic active hepatitis C (hepatitis C virus [HCV]), chronic active hepatitis B (hepatitis B virus [HBV]), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, portal hypertension, or history of autoimmune hepatitis
* Untreated HIV or active hepatitis C detectable by polymerase chain reaction (PCR), or chronic hepatitis B (patients positive for hepatitis B core antibody who are receiving intravenous immunoglobulin therapy [IVIG] are eligible if hepatitis B [HepB] PCR is negative)
* Per PI discretion, active infection that is not well controlled by antibacterial or antiviral therapy

  * Participants with known history of tuberculosis (TB; Mycobacterium tuberculosis) are not eligible for participation. At investigator discretion, latent TB test should be performed for individuals considered to be at high-risk (e.g., immune compromised, persons that have traveled to, or emigrated from, regions with high rates of TB)
* Clinically significant surgery within 2 weeks of enrollment
* Requires use of medications interact with study drug and that cannot be terminated or adjusted. Use of the following therapies requires review by the sponsor investigator:

  * Strong and moderate CYP3A inhibitors
  * Strong and Moderate CYP3A inducers
* Patients with uncontrolled white blood cell count (defined as > 50 K/mm^3 and not controlled with hydroxyurea)
* Patients with known sensitivity to ruxolitinib, venetoclax, or azacitidine
* Since it is unknown whether ruxolitinib, venetoclax, or azacitidine (or their metabolites) are excreted in human milk and because of the potential for serious adverse reactions in the nursing infant, breastfeeding concurrent with study participation is prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) for each arm-specific combination | Up to day 56 (of cycle 1 [cycle length = 28 days]) for non-hematologic DLT and up to day 42 (of cycle 1 [cycle length = 28 days]) for hematologic DLTs
  Within each arm, patient-level toxicity events will be summarized by dose level, major organ category, and grade.

SECONDARY OUTCOMES:
Composite complete remission rate | From first dose to end of cycle 2 (cycle length = 28 days)
  Will be estimated, along with 95% confidence intervals (CIs).
Clinical response rate | From first dose to end of cycle 2 (cycle length = 28 days)
  Will be estimated, along with 95% CIs.
Clinical benefit rate (CBR) | From first dose to end of cycle 2 (up to 36 days)
  CBR will be defined as the proportion of evaluable subjects obtaining stable disease (SD), partial remission, or composite complete remission during the first 2 cycles of therapy. Will be estimated, along with 95% CIs.
Duration of clinical response | From first morphologic leukemia-free state or better to bone marrow blasts >= 5%, circulating blasts, or EMD, or date of last disease assessment, assessed up to 2 years
Duration of clinical benefit | From first SD or better to evidence of progressive disease, or date of last disease assessment, assessed up to 2 years
Event-free survival (EFS) | From first occurrence of treatment failure, disease progression, or death due to any cause, or date of last exam, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method, with median and survival rate estimates at common landmark times reported with 95% log-log CIs. Univariable Cox models will be fit to EFS to assess the impact of baseline patient and disease features; model results such as unadjusted hazard ratios and associated Wald test p-values will be considered hypothesis-generating.
Overall survival (OS) | From date of first dose to death due to any cause or date of last known alive, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method, with median and survival rate estimates at common landmark times reported with 95% log-log CIs. Univariable Cox models will be fit to OS to assess the impact of baseline patient and disease features; model results such as unadjusted hazard ratios and associated Wald test p-values will be considered hypothesis-generating. Median follow-up (and 95% log-log CI) will utilize a patient's OS time and censoring status and be estimated using the reverse Kaplan-Meier method.
Overall incidence of treatment-related and non-treatment related toxicity | From first dose to 30 days after last dose of study agent
  The overall incidence of treatment- related and non-treatment- related toxicity will be determined using the safety-evaluable population. The point estimate and 95% CI for the proportion of patients with each of these toxicity types will be reported. adverse event and abnormal concerning laboratory values will be tabulated by patient and by toxicity event (there can be > 1 event patient) will be tabulated overall and within dose level and summarized by major organ site and severity according to the Common Terminology Criteria for Adverse Events version 5.0.
Changes in patient reported quality of life (QOL) outcomes (Arm 2) | From first dose of study treatment to date of last completed survey, assessed up to 2 years
  Will be assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 and Patient Reported Outcomes Measurement Information System-Fatigue-Short Form 7A. Will be reported with descriptive statistics (e.g., sample size, median, and range) for each survey time point during the treatment period and for (within-patient) changes from baseline. The QOL summary statistics from each survey will be compared to other studies conducted in relapsed/refractory acute myeloid leukemia patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N. Saultz, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided